CLINICAL TRIAL: NCT02290171
Title: Promoting Health in Healthy Living Centres - a Clinical Study Among Famililies With Overweight Children
Brief Title: Promoting Health in Healthy Living Centres - a Clinical Study Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eivind Meland (Other)
Collaborators: University of Agder (Other)
Responsible Party: Sponsor-Investigator, Eivind Meland, Professor, University of Bergen
Organization: University of Bergen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCT02290171
Record Dates: First submitted 2014-10-26; First posted 2014-11-13 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): The intervention groups start the intervention 6 months ahead of the control group.
  Interventions: Behavioral: Activity groups; Behavioral: Group based dietary counselling; Behavioral: Individual counselling
- Delayed intervention group (No Intervention): The control groups will start intervention with 6 months delay

INTERVENTIONS:
Behavioral: Activity groups — Children attend to activity groups weekly during the intervention periode.
  Arms: Intervention group
Behavioral: Group based dietary counselling — Parents attend to four sessions of group based dietary counselling
  Arms: Intervention group
Behavioral: Individual counselling — Parents attend to individual counselling focusing on parental skills and family structure
  Arms: Intervention group

SUMMARY:
The overall aim is to evaluate if a familybased intervention, targeting overweight and obese children and their parents, has a long-term positive effect on weight development and health of the children. The alternative hypothesis to the zero hypothesis is that the children with overweight and obesity who participate in a one-year intervention together with their parents, both at completion of the six months intervention and at long term follow up will have reduced their BMI-for-age z-score (Iso-BMI) and have adopted healthy habits. The behavioral models and educational strategies will be tailored (by age, gender etc.) and include both general information and practical learning sessions.

DETAILED DESCRIPTION:
The investigators intend to perform a controlled clinical trial on interventions on a systemic level.

The target group is overweight and obese children between 6 and 10 years old, their parents, community administrators and public health nurses. The overall aim is to evaluate if a familybased intervention, targeting overweight and obese children and their parents, has a long-term positive effect on weight development of the children. The alternative hypothesis to the zero hypothesis is that the children with overweight and obesity who participate with their parents, both at completion of the six months intervention and at long term follow up (2 years) will have reduced their BMI-for-age z-score (Iso-BMI). The behavioral models and educational strategies will be tailored (by age, gender etc.) and include both general information and practical learning sessions. The program will offer guided active play, defined as spontaneous gross locomotor movement in which children engage to amuse and to occupy themselves.

Parents will attend to workshops intending to increase knowledge and awareness of family structure, healthy eating habits and practical suggestions for implementing healthy behaviors into everyday life. Parents will be educated on how to use these strategies at home, to further support their children in improving their behaviors. This community based study is the support by the local leadership and collaboration with locally based sports clubs. The primary outcome variable, child BMI-for-age z-score will be measured at referral, inclusion, after 6 months, and at 1 and 2 years post intervention. Secondary outcome variables, measured at inclusion and at the end of intervention, are child activity pattern, screen viewing time, eating habits, sleeping patterns and body composition as well as parent BMI, body composition, exercise habits, perception of health, experience of parenthood and level of parental stress.

Physical activity level as well as sleep duration and -quality will be recorded using biaxial accellerometers. A validated food diary will be used. The participants will also be asked to complete a questionnaire including questions about screen viewing time, self-perceived healt, sleeping patterns (children) and perceived autonomy support and autonomous regulations (parents).

ELIGIBILITY:
Inclusion Criteria:

* Iso-BMI>25,
* able to participate in activity groups

Exclusion Criteria:

* Children being unable to participate in activity groups,
* parents not able to participate in group based and individual counseling

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Iso-BMI | Change at 6 months, 1 year, 2 years
  Measure change at 6 month controlled study, and at 1 and 2 years to measure long-term effects

SECONDARY OUTCOMES:
Physical activity level | 6 months, 1 and 2 years
  Measure at the end of the 6 month controlled study, and at 1 and 2 years to measure long-term effects. We will use SenseWear bi-axial accelerometer to mesa sure physics activity.
Dietary habits | 6 months, 1 and 2 years
  Measure at the end of the 6 month controlled study, and at 1 and 2 years to measure long-term effects. We will use a specially designed questionnaire to measure dietary habits.
Self-perceived health | 6 months, 1 and 2 years
  Measure at the end of the 6 month controlled study, and at 1 and 2 years to measure long-term effects. We will use KidScreen 10 questionnaire to measure self-perceived health.

OTHER OUTCOMES:
Autonomous regulation and perceived autonomy support | 6 months, 1 and 2 years
  Measure at the end of the 6 month controlled study, and at 1 and 2 years to measure long-term effects. We will use Treatment Self-regulation Questionnaire to measure autonomous regulation, and Healt Care Climate Questionnaire to measure autonomy support.
Motor skills | 6 months, 1 and 2 years
  Measure at the end of the 6 month controlled study, and at 1 and 2 years to measure long-term effects. We will use Kôrper-koordinationstest fur Kinder to measure motor skills.

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Meland, MD, PhD, Principal Investigator — Dept of Glob Publ Health and Primary Care, University of Bergen
Locations (2):
- Norway (2):
  - University of Bergen, Bergen, Hordaland
  - University of Agder, Kristiansand, Vest-Agder

REFERENCES:
- [Derived] Stea TH, Vettore MV, Ovrebo B, Abildsnes E. Changes in dietary habits and BMI z-score after a 6-month non-randomized cluster-controlled trial among 6-12 years old overweight and obese Norwegian children. Food Nutr Res. 2023 Dec 12;67. doi: 10.29219/fnr.v67.9617. eCollection 2023. PMID 38187797